CLINICAL TRIAL: NCT02320344
Title: Partnerships to Improve Lifestyle Interventions (PILI) 'Ohana Dissemination Project Partners in Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: Kula No Na Po'e Hawaii (Other); Ke Ola Mamo (Other); Hawai'i Maoli (Other); Kokua Kalihi Valley (Unknown)
Responsible Party: Principal Investigator, Joseph Keawe'aimoku Kaholokula, Professor and Chair, University of Hawaii
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MD001660 - PIC
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2017-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (1):
- Partners in Care (Experimental)
  Interventions: Behavioral: Partners in Care

INTERVENTIONS:
Behavioral: Partners in Care — The diabetes self-management intervention is titled, "Partners in Care," emphasizing that there are many individuals and groups that one can call upon to assist with managing one's diabetes. The content includes practical behavioral strategies to improve diabetes self-management practices. The 12 week curriculum provides a basic overview of diabetes and self-management activities, standards of care recommended by the American Diabetes Association, strategies to improve patient-provider communication, support needed for diabetes self-management, information about diabetes medications, and ways to avoid diabetes-related complications.

SUMMARY:
The 3-month face-to-face Partners in Care intervention will be community-based and community-led by trained community peer educators from these four partnering community organizations. The intervention involves 12 weekly, group lessons with each lesson lasting about 1 and 1/2 hours. Individuals with a hemoglobin A1c (HbA1c; average blood sugar levels) greater than or equal to 7% will be recruited for the study because they represent the most at-risk for diabetes-related complications. Over a 3-year accrual period, the community partners will recruit and enroll 150 eligible NHs and PPs, as well as deliver and evaluate the intervention in their respective community settings. The primary outcomes of our study are hemoglobin A1c and self-reported diabetes specific quality of life. Secondary outcomes are cholesterol levels (including HDL, LDL, total cholesterol, and triglycerides), blood pressure, body mass index, and psychosocial adaptation.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age >18 years of age,
2. English-speaking,
3. Physician-diagnosed type 2 diabetes, and
4. Baseline hemoglobin A1c >7%.

Exclusion Criteria:

1. Survival less than 6 months,
2. Planning to move out of the community during the intervention study period,
3. Pregnancy,
4. Any co-morbid condition (physical and mental disabilities) that would prevent the individual from participating in the intervention protocol (i.e., major psychiatric illness).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-07; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 3 months
  change in hemoglobin A1c from baseline to 3-months
Problem Areas in Diabetes | 3 months
  The Problem Areas in Diabetes (PAID) will be used to assess diabetes specific quality of life. Change in PAID score from baseline to 3-months

SECONDARY OUTCOMES:
Total Cholesterol (including HDL and LDL) | 3 months
  change in cholesterol from baseline to 3 months
Triglycerides | 3 months
  change in triglycerides from baseline to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Native Hawaiian Health, University of Hawaii, Honolulu, Hawaii, United States